CLINICAL TRIAL: NCT04061863
Title: A Phase IB/II, Single Arm, Multi-center Study of Nivolumab in Combination With Eribulin in HER2 Negative Metastatic Breast Cancer Patients
Brief Title: Nivolumab and Eribulin in HER2 Negative Metastatic Breast Cancer
Acronym: KORNELIA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Korean Cancer Study Group (KCSG) (Unknown); Eisai Korea Inc. (Industry); Ono pharmaceutical Korea (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCSG BR18-16
Record Dates: First submitted 2019-08-13; First posted 2019-08-20 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; eribulin; nivolumab; immunotherapy; immune checkpoint inhibitor; metastatic breast cancer; PD-1
MeSH Terms: conditions — Breast Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: ER+/HER2- BC cohort: 45 pts ER-/HER2- (Triple negative) BC cohort: 45 pts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ER+/HER2- breast cancer (Experimental): will be treated with a combination of eribulin and nivolumab
  Interventions: Drug: Nivolumab
- ER-/HER2- breast cancer (Experimental): will be treated with a combination of eribulin and nivolumab
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 360mg on D1 every 3 weeks Eribulin 1.4mg/m2 on D1, 8 every 3 weeks
  Other Names: Opdivo

SUMMARY:
Cancer therapeutics such as chemotherapy may modulate tumor/immune-system interactions in favor of the immune system. Chemotherapy can result in tumor cell death with a resultant increase in tumor antigen delivery to antigen-presenting cells. Therefore, combining immunotherapy (Nivolumab) with chemotherapy (Eribulin) is a promising anti-cancer strategy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Age 20 years or older
* ECOG performance status(PS) 0 or 1
* Histologically confirmed stage IV or recurrent breast cancer
* HER2 negative disease: not eligible for anti-HER2 therapy

  * HER2 negative [IHC 0, 1+ or IHC 2+ with corresponding ISH non-amplified or ratio less than 2.0 or ISH non-amplified ratio less than 2.0] as per ASCO-CAP HER2 guideline recommendations 2013 (ASCO-CAP)
* Patients previously treated with anthracycline and/or taxane unless contraindicated; Patients who received anthracycline and/or taxane based chemotherapy in either the neoadjuvant, adjuvant or metastatic setting and experienced disease progression on or after taxane-based chemotherapy in the metastatic setting
* No more than 3 prior lines of cytotoxic chemotherapy for metastatic disease; patients who experienced disease recurrence within 1 year after completion of (neo)adjuvant anthracycline and taxane-based chemotherapy will be counted as 1 prior line of treatment.; hormonal therapy will not be counted as a prior line of treatment
* Measurable disease according to RECIST v 1.1.

Exclusion Criteria:

* Previous treatment with eribulin mesylate or any anti-PD-1, PD-L1, or PD-L2
* Active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment.
* Known central nervous system (CNS) disease, except for those subjects with treated brain metastasis who are stable for at least 1 month, having no evidence of progression or hemorrhage after treatment and no ongoing requirement for corticosteroids, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]) during the screening period
* Known history of human immunodeficiency virus (HIV) positive
* Known active hepatitis B or hepatitis C (eg, HCV RNA detected)
* Any other malignancy that required treatment or has shown evidence of recurrence (except for nonmelanoma skin cancer, or histologically confirmed complete excision of carcinoma in situ) during the 3 years prior to enrollment in this study
* History of significant cardiovascular disease
* Hypersensitivity to the active substance or any other excipients of the eribulin mesylate drug product, or to nivolumab
* Scheduled for major surgery during the study
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be allowed
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has a history of interstitial lung disease
* Has received a live-virus vaccination within 30 days of planned start of study therapy. Seasonal flu vaccines that do not contain live virus are permitted.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
6 months progression-free survival (PFS) rate | 6 months

SECONDARY OUTCOMES:
Objective response rate by RECIST criteria v 1.1 | 2 years
Overall survival (OS) | 2 years (upto 5 years)
Incidence Rate of each Toxicity by CTCAE 4.0 | 2 years (upto 5 years)
Clinical benefit rate by RECIST criteria v 1.1 (and iRECIST) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: JEEHYUN KIM, MD,PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park C, Suh KJ, Kim SH, Lee KH, Im SA, Kim MH, Sohn J, Jeong JH, Jung KH, Lee KE, Park YH, Kim HJ, Cho EK, Choi IS, Noh SJ, Shin I, Cho DY, Kim JH. Genomic and transcriptomic profiles associated with response to eribulin and nivolumab combination in HER-2-negative metastatic breast cancer. Cancer Immunol Immunother. 2024 Aug 6;73(10):197. doi: 10.1007/s00262-024-03782-7. PMID 39105849
- [Derived] Kim SH, Im SA, Suh KJ, Lee KH, Kim MH, Sohn J, Park YH, Kim JY, Jeong JH, Lee KE, Choi IS, Park KH, Kim HJ, Cho EK, Park SY, Kim M, Kim JH. Clinical activity of nivolumab in combination with eribulin in HER2-negative metastatic breast cancer: A phase IB/II study (KCSG BR18-16). Eur J Cancer. 2023 Dec;195:113386. doi: 10.1016/j.ejca.2023.113386. Epub 2023 Oct 14. PMID 37890351
- See also: Korea Cancer Study Group — https://www.kcsg.org/en/index.do
- See also: Seoul National University Bundang Hospital — https://www.snubh.org/index.do